CLINICAL TRIAL: NCT01110707
Title: Lutropin Alpha in the Middle of the Controlled Ovarian Stimulation Follicular Phase in Women With Reduced Ovarian Reserve: Comparative Study, in Phase II, With Parallel Control
Brief Title: A Randomised, Phase II, Comparative Study With a Parallel Control for Evaluating the Efficacy and Safety of Combined Treatment of Lutropin Alpha and Recombinant Human Luteinizing Hormone in the Middle of the Controlled Ovarian Stimulation Follicular Phase in Women With Reduced Ovarian Reserve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP 25186
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2017-08

CONDITIONS: Infertility; Ovulation Induction
Keywords: Reproductive technology, Assisted; Recombinant human follicle stimulating hormone (r-hFSH); Recombinant leutinizing hormone (r-hLH); Ovulation induction; Infertility
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa; Luteinizing Hormone, beta Subunit

ARMS (2):
- r-hFSH + r-hLH (Experimental)
  Interventions: Drug: Recombinant human follicle stimulating hormone (r-hFSH); Drug: Recombinant human luteinizing hormone (r-hLH)
- r-hFSH alone (Active Comparator)
  Interventions: Drug: Recombinant human luteinizing hormone (r-hLH)

INTERVENTIONS:
Drug: Recombinant human follicle stimulating hormone (r-hFSH) — Subjects will receive subcutaneous injection of recombinant human follicular stimulating hormone (r-hFSH) 300-450 International Units (IU) administered after pituitary desensitization according to the ovarian response with gonadotrophin-releasing hormone agonist (GnRH-a; at a dose of 0.1 milligram per day [mg/day]).
  Other Names: GONAL-f; Follitrophin alpha
  Arms: r-hFSH + r-hLH
Drug: Recombinant human luteinizing hormone (r-hLH) — Subjects will receive subcutaneous injection of recombinant human luteinizing hormone (r-hLH) 150 IU/day until the end of ovarian stimulation.
  Other Names: Luveris; Lutrophin alpha

SUMMARY:
This was a prospective, randomized, Phase II, comparative study with a parallel control for evaluating the efficacy and safety of combined treatment of recombinant human follicle stimulating hormone (r-hFSH) and recombinant human luteinizing hormone (r-hLH). The combined treatment was administered at the middle of the follicular phase in subjects undergoing in-vitro fertilisation (IVF) through intracytoplasmic sperm injection (ICSI) and transfer of embryos (ET).

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following inclusion criteria within the 6 months prior to starting the pituitary suppression unless otherwise specified:

* Postmenopausal woman aged between 35 and 40 years that wishes to become pregnant
* Subjects with basal serum level (beginning of the follicular phase, Day 2-5) of Follicle-Stimulating Hormone (FSH) less than 10 IU/L determined within the 6 months prior as well as Luteinizing hormone (LH) and Estradiol (E2) levels within the normal interval according to standard data for the area where the study was carried out
* Subjects with a regular menstrual cycles between 25-35 days
* Subjects with infertility that justifies treatment with IVF/ET or ICSI
* Subjects undergoing controlled ovarian stimulation (COS) with r-hFSH using a long protocol with GnRH-a
* Sperm availability from the subject's current partner unless it is planned to use sperm from a donor
* Subjects with both ovaries
* Subjects with uterine cavity capable of withstanding the implantation of the embryo and pregnancy
* Subjects whose vaginal smear (PAP) was normal within the 3 years prior to starting the stimulation
* Subjects with body mass index (BMI) between 18 and 30 at the time of participation in the study
* Subjects in whom at least 30 days have elapsed since the last dose of clomiphene citrate or gonadotropins before beginning treatment with GnRH-a
* Subjects with a negative pregnancy test result using the beta human chorionic gonadotropin (beta-hCG) test (in urine or blood) before beginning treatment with GnRH-a
* Subjects willing to and capable of following the protocol during the entire study
* Subjects who have provided informed written consent before carrying out any procedure related with the study (that is not part of the normal medical treatment followed by the subject)

Exclusion Criteria:

* Subject who were human immunodeficiency virus, hepatitis B and C virus positive
* Subjects suffering from any clinically important systematic disease, hypothalmic or pituitary tumour, ovarian, uterine or breast cancer, endocrinopathy and/or medical alterations, biochemical or hematological that as per the investigators judgement, may interfere with the gonadotropin treatment
* Subjects who have been subjected to more than 2 assisted reproductive cycles in the past
* Subjects who have cancelled 2 cycles in the past
* Subjects who have cryopreserved embryos from previous assisted reproductive cycles
* Subjects with non explained vaginal haemorrhages
* Subjects with polycystic ovary, enlarged ovary or ovarian cysts of unknown aetiology
* Subjects with any contraindication for getting pregnant or taking the pregnancy to full term
* Subjects with known allergy to the gonadotropin preparations or any of its excipients
* Subjects with current drug use or prior personal history of alcohol, drug or psychiatric drug dependency in the past five years
* Subjects with prior participation in this study or simultaneous participation in a different clinical study with a medication under investigation
* Subjects who were not willing to or incapable of following the study protocol

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2005-01-10 (Actual); Primary Completion 2006-11-15 (Actual); Study Completion 2006-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Hospital de Cruces, Plaza de Cruces, 12, 48903, Vizcaya, Spain

REFERENCES:
- [Result] Matorras R, Prieto B, Exposito A, Mendoza R, Crisol L, Herranz P, Burgues S. Mid-follicular LH supplementation in women aged 35-39 years undergoing ICSI cycles: a randomized controlled study. Reprod Biomed Online. 2009 Dec;19(6):879-87. doi: 10.1016/j.rbmo.2009.09.016. PMID 20031032
- [Result] Matorras R, Prieto B, Exposito A, Mendoza R, Crisol L, Herranz P, Burgues S. Mid-follicular LH supplementation in women aged 35-39 years undergoing ICSI cycles: a randomized controlled study. Reprod Biomed Online. 2011 Feb;22 Suppl 1:S43-51. doi: 10.1016/S1472-6483(11)60008-4. PMID 21575849

RESULTS

PARTICIPANT FLOW:
Groups:
- r-hFSH + r-hLH: Subjects received subcutaneous injection of recombinant human follicular stimulating hormone (r-hFSH) 300-450 International Units (IU) administered after pituitary desensitization according to the ovarian response with gonadotrophin-releasing hormone agonist (GnRH-a; at a dose of 0.1 milligram per day [mg/day]) along with subcutaneous injection of recombinant human luteinizing hormone (r-hLH) 150 IU/day until the end of ovarian stimulation. Administration of both r-hFSH and r-hLH was suspended 36 hours before administering recombinant human chorionic gonadotrophin (r-hCG).
- r-hFSH Alone: Subjects received subcutaneous injection of a recombinant human follicular stimulating hormone (r-hFSH) 300-450 International Units (IU) administered after pituitary desensitization according to the ovarian response with gonadotrophin-releasing hormone agonist (GnRH-a; at a dose of 0.1 milligram per day [mg/day]).
Period: Overall Study
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Started | 63 | 68
Completed | 63 | 65
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone | Total
Number analyzed (Participants) | 63 | 68 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 68 | 131
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 68 | 131
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Metaphase II (M-II) Oocytes Retrieved
Description: Mean number of M-II oocytes were calculated for subjects undergoing ovum pick up for Intra-cytoplasmic Sperm Injection (ICSI). ICSI is an in-vitro fertilization procedure in which a single sperm is injected directly into an egg under a microscope. Metaphase II stage of the oocyte was classified as the time at which the first polar body was observed microscopically. Metaphase II oocytes are a sub-group of the total number of oocytes.
Time Frame: 36 hours post r-hCG administration
Population: The Intention-To-Treat (ITT) analysis set included all the randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: M-II oocytes
Groups:
- r-hFSH + r-hLH: GONAL-f (follitropin alpha); a recombinant human follicular stimulating hormone (r-hFSH) injection 300-450 International Units (IU) subcutaneously (SC) was administered separately after achieving pituitary desensitization according to the ovarian response with gonadotrophin-releasing hormone agonist (GnRH-a) at a dose of 0.1 milligram per day (mg/day). Subjects also received Luveris; recombinant human luteinizing hormone (r-hLH) injection 150 IU/day SC until the end of ovarian stimulation. Administration of both r-hFSH and r-hLH was suspended 36 hours before administering recombinant human chorionic gonadotrophin (r-hCG).
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
M-II oocytes | 6.7 (4.1) | 7.0 (4.8)

2. Secondary Outcome: Number of Fertilized Oocytes (2 Pronuclei [2PN])
Description: Oocytes were fertilized using Intra-cytoplasmic Sperm Injection (ICSI) technique which is an in-vitro fertilization procedure in which a single sperm is injected directly into an egg under a microscope. The appearance of 2PN is the first sign of successful fertilization as observed during in vitro fertilization, and is usually observed after ICSI. The zygote is then termed 2PN.
Time Frame: 36 hours post r-hCG administration
Population: The ITT analysis set included all the randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: 2PN oocytes
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
2PN oocytes | 3.1 (2.3) | 3.3 (2.6)

3. Secondary Outcome: Quality of Embryos
Description: Embryos were classified into 5 different grades (1 to 5) based on their capacity of implantation. Grade 1 embryos were those with best capacity of implantation and Grade 5 embryos were those with worst capacity of implantation. Mean number of embryos for each of the 5 grades were reported.
Time Frame: Day 2-3 post r-hCG administration
Population: The ITT analysis set included all the randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
embryos
  Grade 1 | 1.1 (1.1) | 1.3 (1.4)
  Grade 2 | 1.1 (1.5) | 1.2 (1.1)
  Grade 3 | 0.5 (0.6) | 0.5 (0.9)
  Grade 4 | 0.3 (0.5) | 0.2 (0.6)
  Grade 5 | 0.3 (1.0) | 0.2 (0.6)

4. Secondary Outcome: Embryo Implantation Rate
Description: Embryo implantation rate was measured as the number of gestational sacs observed divided by the number of embryos transferred multiplied by 100.
Time Frame: 35-42 days post r-hCG administration
Population: The ITT analysis set included all the randomized subjects who received at least 1 dose of study medication.
Measure: Number; unit: Percent sacs per embryo
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
Percent sacs per embryo | 18.1 | 11.3

5. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy rate defined as the percentage of subjects with a ultrasound confirmation of a gestational sac, with or without fetal heart activity.
Time Frame: 35-42 days post r-hCG administration
Population: The ITT analysis set included all the randomized subjects who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of subjects
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
Percentage of subjects | 27.0 | 14.7

6. Secondary Outcome: Mean Number of Follicles Greater Than or Equal to (>=) 14 Millimeter (mm)
Description: Mean number of follicles as per the following categories were presented: >=14 mm and less than (<) 16 mm; >=16 mm and <18 mm and >=18 mm.
Time Frame: r-hCG day (end of stimulation cycle [approximately 28 days])
Population: The ITT analysis included all the randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
Follicles
  >=14 mm and <16 mm | 2.2 (2.0) | 2.1 (1.9)
  >=16 mm and <18 mm | 2.3 (2.0) | 2.7 (2.1)
  >=18 mm | 4.0 (3.0) | 3.7 (3.0)

7. Secondary Outcome: Endometrial Thickness
Time Frame: r-hCG day (end of stimulation cycle [approximately 28 days])
Population: The ITT analysis set included all the randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
mm | 6.0 (3.2) | 5.9 (3.2)

8. Secondary Outcome: Number of Cycles Cancelled Due to Unsatisfactory Response
Description: If the subject was not administered with r-hCG and withdrew prematurely from the trail, it is considered as cycle cancellation
Time Frame: r-hCG day (end of stimulation cycle [approximately 28 days])
Population: The ITT analysis included all the randomized subjects who received at least one dose of study medication.
Measure: Number; unit: cycles
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
cycles | 0 | 3

9. Secondary Outcome: Mean Number of Oocytes Retrieved
Description: Oocyte retrieval is a technique used in in-vitro fertilization (IVF) in order to remove oocyte from the ovary of the female subject, enabling fertilization outside the body.
Time Frame: 36 hours post r-hCG administration
Population: The ITT analysis included all the randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Number analyzed (Participants) | 63 | 68
Oocytes | 8.3 (4.7) | 8.9 (4.9)

ADVERSE EVENTS:
Arm/Group | r-hFSH + r-hLH | r-hFSH Alone
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/68
Other Adverse Events (participants affected / at risk) | 2/63 | 0/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | r-hFSH + r-hLH (N=63) | r-hFSH Alone (N=68)
Ovarian Hyperstimulation Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pelvic Inflammatory Disease (Pregnancy, puerperium and perinatal conditions) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other